CLINICAL TRIAL: NCT01131273
Title: Suboxone and Methadone for HIV Risk Reduction in Subutex Injectors
Brief Title: HIV Risk Reduction in Subutex Injectors in Tbilisi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDA026754A; R21DA026754 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2010-04-08; First posted 2010-05-26 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: HIV
Keywords: buprenorphine injecting; opiate dependence; HIV risk; treatment outcome; opiate dependence with buprenorphine injecting
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone; Buprenorphine, Naloxone Drug Combination; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone maintenance for 12 weeks (Active Comparator): Methadone maintenance for 12 weeks as compared to 12 weeks maintenance on Suboxone.
  Interventions: Drug: methadone
- buprenorphine-naloxone (Suboxone) (Active Comparator): 12 weeks of maintenance on buprenorphine-naloxone (Suboxone) at daily doses ranging from 8 to 32 mg with counseling
  Interventions: Drug: buprenorphine-naloxone (Suboxone) for 12 weeks

INTERVENTIONS:
Drug: methadone — 12 weeks of methadone maintenance with counseling
  Arms: Methadone maintenance for 12 weeks
Drug: buprenorphine-naloxone (Suboxone) for 12 weeks — 12 weeks of maintenance with counseling
  Arms: buprenorphine-naloxone (Suboxone)

SUMMARY:
This study will obtain pilot data on the acceptability of a 12-week course of daily observed suboxone and methadone, followed by a dose taper or referral to a local treatment program for 80 opioid dependent patients (40 group) who have been injecting subutex or other buprenorphine preparations 10 or more days in the past 30, and on the impact of each medication on HIV risk and on subutex and opioid use during treatment and a followup at week 20. it will be done at the Uranti Methadone Program, affiliated with the Addiction Research Center, Union Alternative of Georgia in Tbilisi.

ELIGIBILITY:
Inclusion Criteria:

* current opioid dependence;
* injecting buprenorphine 10 or more times in the last 30 days;
* between 25 and 50 years of age;
* buprenorphine and/or opiate positive urine test;
* not on methadone maintenance in last 4 weeks;
* stable address within Tbilisi and not planning to move;
* home or cellular phone number where can be reached;
* able to provide name of family member who knows whereabouts;
* willingness and ability to give informed consent.

Exclusion Criteria:

* currently dependent on alcohol, benzodiazepines or other CNS depressants;
* legan charges with impending incarceration;
* plans to move from Tbilisi within next 6 months;
* current participation in another treatment study;
* serious medical problems that would impair or make hazardous ability to participate;
* active TB;
* currently psychotic/suicidal;
* uncontrolled seizure disorder.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2010-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Buprenorphine injecting | 12 weeks
  1) Obtain pilot data on the impact of a 12-week course of daily, observed Suboxone and methadone treatment on HIV injecting risk behavior, particularly that associated with injecting use of Subutex. 2) obtain pilot data on the degree to which the target population accepts treatment with daily observed Suboxone and methadone.

SECONDARY OUTCOMES:
HIV Risk | 12 weeks
  Obtain pilot data on the degree to which a 12-week course of suboxone or methadone reduces illegal activities and improves employment, psychiatric symptoms, overall adjustment and assess the prevalence of HIV, HEP B/C among study patients at week 20.

CONTACTS AND LOCATIONS:
Overall Officials: Geroge Woody, MD, Study Director — University of Pennsylvania
Locations (1):
- Union Alternative Georgia, Tbilisi, Georgia

REFERENCES:
- [Derived] Otiashvili D, Piralishvili G, Sikharulidze Z, Kamkamidze G, Poole S, Woody GE. Methadone and buprenorphine-naloxone are effective in reducing illicit buprenorphine and other opioid use, and reducing HIV risk behavior--outcomes of a randomized trial. Drug Alcohol Depend. 2013 Dec 1;133(2):376-82. doi: 10.1016/j.drugalcdep.2013.06.024. Epub 2013 Jul 31. PMID 23916321